CLINICAL TRIAL: NCT01522690
Title: Assessment of Accelerometric Measurement Devices for Gait Analysis
Acronym: ACCELERIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Myologie, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ACCELERIX
Record Dates: First submitted 2012-01-04; First posted 2012-02-01 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: Accelerometer; gait analysis; Healthy subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Different walk tests with an accelerometer device — Subjects will performed three walk tests of 50 meter at different speeds, a six minute walk test, a walking test of 30 seconds then a test to measure the maximum force of extension and knee flexion on each leg. The walk tests will be performed with the accelerometer device (Locometrix) worn in a belt

SUMMARY:
The objective of this study is to obtain normative accelerometry data during the six minute walk test and a 30 second walk test on healthy subjects in order to determine the accelerometric variables that are the most relevant to describe gait disorders in patient populations. Secondary objectives of this study are to investigate the impact of walking speed and muscle strength on the accelerometric parameters, to assess the reproducibility of the method and to compare accelerometric data obtained with two different devices.

ELIGIBILITY:
Inclusion Criteria:

* healthy ambulant subject
* subject affiliated to a social security system
* subject who signed an informed consent

Exclusion Criteria:

* surgery or recent trauma to the lower limbs (under 6 months)
* high performance sport
* chronic treatment alters the strength in the month before inclusion
* pregnant or nursing woman
* person under guardianship or curatorship
* orthopedic, neuromuscular or neurological disease having an impact on the quality of walking

Ages: 5 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Accelerometric variables measured for each walk test | At baseline
Accelerometric variables measured for each walk test | 1 hour after baseline

SECONDARY OUTCOMES:
Gait speed measured for each walk test | At baseline
Knee flexion and extension strength | At baseline
Gait speed measured for each walk test | 1 hour after baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Myologie - GH Pitié Salpêtrière, Paris, Paris, France